CLINICAL TRIAL: NCT00339846
Title: Genetic Analysis of Craniofrontonasal Syndrome
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905029; 05-HG-N029
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-09-17

CONDITIONS: Craniofrontonasal Syndrome; CFNS
Keywords: Craniosynostosis; Craniofrontonasal Syndrome; CFNS
MeSH Terms: conditions — Craniofrontonasal dysplasia; Craniosynostoses

SUMMARY:
This study will determine whether all patients with craniofrontonasal syndrome (CFNS) have a mutation of a gene called ephrin-B1 (EFNB1). CFNS is one of a group of conditions called craniosynostosis syndromes that result from closure of one or more of the fibrous joints between the bones of the skull before brain growth is complete. Because of the premature closure, the brain is not able to grow in its natural shape; instead, there is growth in areas of the skull where the joints have not yet closed. In CFNS, it results in malformation of the skull and face. It is known that the EFNB1 mutation can cause CFNS, and this study will see if the gene change is present in all patients with the disorder.

This study includes patients and family members affected with CFNS. Participants have 1 to 2 teaspoons of blood drawn for genetic studies. A second blood sample may be requested for further research. Some blood may be used to establish a cell line for later studies. This involves growing the white blood cells from the blood sample. The cells can be kept in the laboratory to make more DNA or can be frozen for later use in studies of craniosynostosis. Patients may also have their medical records reviewed to relate gene changes to clinical features in CFNS.

DETAILED DESCRIPTION:
The scientific objective of this study is to determine if all patients with Craniofrontonasal Syndrome (CFNS) contain mutations in the ephrin-B1 (EFNB1) gene in Xq12. We will use mutational analysis of EFNB1 as our principal tool to study the genetics of CFNS. Previously, we had mapped the CFNS locus to a 13 cM region in Xp22 using linkage analysis of 12 unrelated CFNS families with 2 or more affected family members in 2-4 generations. More recently there have been two reports that 23 independent CFNS patients all have mutations in the EFNB1 located at Xq12. Hence, either CFNS displays genetic heterogeneity with at least two genes (one in Xp22 and EFNB1) or our previous linkage analysis was inaccurate and all CFNS patients have EFNB1 mutations.

We have previously collected a large number of coded blood samples from patients with DFNS. We propose to sequence the EFNB1 in all 12 of our previously published CFNS families as well as 6 additional families, 22 sporadic CFNS patients, and two CFNS patients with chromosomal anomalies.

We will be sending letters to all physicians who have referred CFNS patients to us in the past for molecular studies. This letter will outline the recent developments identifying EFNB1 as the CFNS gene. We would like to utilize the referring physicians as liaisons between our lab and CFNS patients. Through the referring physicians, we will invite the patients and their families to join a new study if they are interested in obtaining their genetic testing results. All of our results will be confirmed by a CLIA-certified lab prior to being given to patients or referring physicians.

ELIGIBILITY:
* INCLUSION CRITERIA:

CFNS patients and their families who were previously referred to us; the majority have DNA samples and clinical data already archived in our collection.

EXCLUSION CRITERIA:

Anyone unwilling to provide informed consent (for themselves as adults, or on behalf of their children as minors) or assent.

We generally reviewed a brief clinical description from the referring physician about a potential research subject to determine that the subject was appropriate to enter into the study. We reserved the right to exclude cases that were clearly not related to our direct research interests.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152
Dates: Start 2005-01-05; Study Completion 2008-09-17

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Hospital, Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Compagni A, Logan M, Klein R, Adams RH. Control of skeletal patterning by ephrinB1-EphB interactions. Dev Cell. 2003 Aug;5(2):217-30. doi: 10.1016/s1534-5807(03)00198-9. PMID 12919674
- [Background] Davy A, Aubin J, Soriano P. Ephrin-B1 forward and reverse signaling are required during mouse development. Genes Dev. 2004 Mar 1;18(5):572-83. doi: 10.1101/gad.1171704. PMID 15037550
- [Background] Feldman GJ, Ward DE, Lajeunie-Renier E, Saavedra D, Robin NH, Proud V, Robb LJ, Der Kaloustian V, Carey JC, Cohen MM Jr, Cormier V, Munnich A, Zackai EH, Wilkie AO, Price RA, Muenke M. A novel phenotypic pattern in X-linked inheritance: craniofrontonasal syndrome maps to Xp22. Hum Mol Genet. 1997 Oct;6(11):1937-41. doi: 10.1093/hmg/6.11.1937. PMID 9302274